CLINICAL TRIAL: NCT06032598
Title: Clinical-instrumental Evaluation of the Efficacy of Two Dietary Supplements Claiming Anti-aging Properties and Skin Complexion Improvement. A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Evaluation of the Anti-aging Efficacy of Two Dietary Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0003588/23
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Berry extract 1 (Experimental): Dietary supplement - Berry extract 1
  Interventions: Dietary Supplement: Berry extract 1
- Berry extract 2 (Experimental): Dietary supplement - Berry extract 2
  Interventions: Dietary Supplement: Berry extract 2
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Berry extract 1 — The study foresees the intake of 1 capsule per day during 84 days
  Arms: Berry extract 1
Dietary Supplement: Berry extract 2 — The study foresees the intake of 1 capsule per day during 84 days
  Arms: Berry extract 2
Dietary Supplement: Placebo — The study foresees the intake of 1 capsule per day during 84 days
  Arms: Placebo

SUMMARY:
The study is aimed to assess the efficacy of two dietary supplements composed of berry extracts in reducing skin aging signs and improving skin complexion.

DETAILED DESCRIPTION:
A double blind, parallel groups, placebo-controlled study is carried out on 90 healthy female subjects aged between 35 and 65 (±2) years old with phototypes from I to III, uneven skin tone, visible Crow's feet wrinkles and mild-moderate skin slackness at cheek level.

The study foresees 84 days of products intake. Evaluations of the parameters under study are performed at baseline, after 28, 56 and 84 days of products consumption.

ELIGIBILITY:
Inclusion criteria :

* Healthy female subjects,
* Caucasian ethnicity,
* Age between 35 and 65 (limits of ±2 years old could be included)
* Phototypes from I to III
* Subject with uneven skin tone (grade 1-3 - internal clinical scale)
* Subject with visible Crow's feet wrinkles (≥2 according to Skin Aging Atlas - Caucasian and Asian Type - Bazin Roland)
* Subject with mild-moderate skin slackness at cheek level (grade 1-3 - internal clinical scale).
* Willingness to not assume during the study period products other than the test product
* Subjects registered with National Health Service (NHS)
* Subjects certifying the truthfulness of the personal data disclosed to the investigator
* Subjects able to understand the language used in the investigation centre and the information given by the investigator
* Subjects able to respect the instructions given by the investigator as well as able to respect the study constraints and specific requirements
* The pharmacological therapy (except for the pharmacological therapy in the non-inclusion criteria) should be stable for at least one month without any changes expected or planned during the study
* Commitment not to change the daily routine or the lifestyle
* Subjects who have not been recently involved in any other similar study (at least one month of wash-out)
* Subject under effective contraception (oral/not oral) therapy
* Subjects who accept not to expose in intensive way to UV rays during the whole study duration.
* Subject aware of the study procedures and having signed an informed consent form and privacy information form.

Exclusion Criteria:

* Subject does not meet the inclusion criteria,
* Subjects with acute or chronic diseases able to interfere with the outcome of the study or that are considered dangerous for the subject or incompatible with the study requirements
* Subjects participating or planning to participate in other clinical trials
* Subjects deprived of freedom by administrative or legal decision or under guardianship
* Subjects not able to be contacted in case of emergency
* Subjects admitted to a health or social facility
* Subjects planning a hospitalisation during the study
* Subjects who participated in a similar study without respecting an adequate washout period
* Subjects having an acute, chronic or progressive illness liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subjects under pharmacological treatments that are considered incompatible with the study requirement by the investigator
* Subjects having a skin disease or condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subject with known or suspected sensitization to one or more test formulation ingredients
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (for the women of childbearing potential)
* Consumption of food supplement(s) and/or use of topical skincare products with whitening activity currently or within the past 4 weeks before the study
* Subjects accustomed to use tanning beds
* Subjects taking medication with photosensitizing potential, drugs and/or dietary supplements able to induce skin coloring, corticoids, currently or during the month before the study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Skin profilometry | Baseline
  Primos 3D
Skin profilometry | 28 days
  Primos 3D
Skin profilometry | 56 days
  Primos 3D
Skin profilometry | 84 days
  Primos 3D

SECONDARY OUTCOMES:
Skin elasticity | Baseline
  Cutometer
Skin elasticity | 28 days
  Cutometer
Skin elasticity | 56 days
  Cutometer
Skin elasticity | 84 days
  Cutometer
Skin color | Baseline
  CIELab color space
Skin color | 28 days
  CIELab color space
Skin color | 56 days
  CIELab color space
Skin color | 84 days
  CIELab color space
Crow's feet | Baseline
  Clinical evaluation (Skin Aging Atlas - Caucasian and Asian Type - Bazin Roland)
Crow's feet | 28 days
  Clinical evaluation (Skin Aging Atlas - Caucasian and Asian Type - Bazin Roland)
Crow's feet | 56 days
  Clinical evaluation (Skin Aging Atlas - Caucasian and Asian Type - Bazin Roland)
Crow's feet | 84 days
  Clinical evaluation (Skin Aging Atlas - Caucasian and Asian Type - Bazin Roland)
Skin firmness | Baseline
  Clinical scoring (internal validated scale from 1 to 5, where: 1 = not firm skin and 5 = very firm skin)
Skin firmness | 28 days
  Clinical scoring (internal validated scale from 1 to 5, where: 1 = not firm skin and 5 = very firm skin)
Skin firmness | 56 days
  Clinical scoring (internal validated scale from 1 to 5, where: 1 = not firm skin and 5 = very firm skin)
Skin firmness | 84 days
  Clinical scoring (internal validated scale from 1 to 5, where: 1 = not firm skin and 5 = very firm skin)
Skin homogeneity improvment from baseline | 28 days
  Clinical scoring (internal validated scale from 1 to 4, where: 1 = no variation and 4 = evident variation)
Skin homogeneity improvment from baseline | 56 days
  Clinical scoring (internal validated scale from 1 to 4, where: 1 = no variation and 4 = evident variation)
Skin homogeneity improvment from baseline | 84 days
  Clinical scoring (internal validated scale from 1 to 4, where: 1 = no variation and 4 = evident variation)
Self-assessment of product efficacy | 84 days
  Questionnaire (20 questions with 4 possible answers : completely agree / agree / disagree / completely disagree)
Skin antioxidant potential | Baseline
  FRAP (Ferric Reducing Antioxidant Power) assay
Skin antioxidant potential | 84 days
  FRAP (Ferric Reducing Antioxidant Power) assay

CONTACTS AND LOCATIONS:
Overall Officials: Ileana De Ponti, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia srl, Milan, Italy